CLINICAL TRIAL: NCT05137158
Title: The Effect of Intermittent Theta Burst Stimulation on Negative Symptoms And Cognitive Function in Schizophrenia
Brief Title: iTBS on Negative Symptoms and Cognitive Function in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WU202110TBS
Record Dates: First submitted 2021-11-09; First posted 2021-11-30 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; iTBS; Negative Symptom; Cognitive function
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Sixty participants are randomly and equally divided into intervention group or sham stimulation group according to the predetermined random number list.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iTBS stimulation (Experimental): The patients in iTBS stimulation group will receive iTBS stimulation on the target of the left dorsolateral prefrontal cortex for 10 consecutive days and 3 times per day.There will have at least 30 minutes interval between each intervention.
  Interventions: Device: Intermittent theta burst stimulation
- Sham stimulation (Sham Comparator): The participants in sham stimulation will receive sham stimulation, as the coil vertical to the brain surface, for 10 consecutive days and 3 times per day.There will have at least 30 minutes interval between each intervention.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Intermittent theta burst stimulation — Intermittent theta burst stimulation(iTBS) on the left DLPFC, the left DLPFC will be targeted utilizing the localite neuronavigation system. The stimulation intensity is set at 80% of resting motor threshold(RMT), and the other parameters are set to triplet 50Hz bursts, repeat at 5Hz, 2s seconds on and 8 seconds off, 600 pulses per session, total duration of 3 minutes and 20 seconds.
  Arms: iTBS stimulation
Device: Sham stimulation — The same procedure will be performed in sham group including the RMT assessment and the neuronavigation system for target localization, but the sham coil will vertical to the brain surface and deliver a very slight magnetic field, which have the same appearance and sound, and provide the same tactile sensations as the active coils.
  Arms: Sham stimulation

SUMMARY:
The negative symptoms and cognitive deficits are common in patients with schizophrenia, and do not respond well to antipsychotics. The effective treatments for negative symptoms and cognitive impairment are still to be explored. rTMS is a safe and non-invasive physical treatment, some studies has been indicated that the high frequency rTMS could increase the excitability of cortex, and has potentials to improve negative symptoms and cognitive function in schizophrenia. In this study, we explore the effects of iTBS on negative symptoms and cognitive function based on identifying the brain network connection of schizophrenia symptoms.

DETAILED DESCRIPTION:
The negative symptoms and cognitive deficits are two core symptoms in patients with schizophrenia, and do not respond well to antipsychotics. There are many researches on the biological mechanism of these two symptoms, and some studies indicated that these two symptoms maybe related to the dysfunction of prefrontal cortex and deficiency of dopamine. rTMS is a safe and non-invasive physical treatment, some studies has been indicated that the high frequency rTMS could increase the excitability of cortex, and has potentials to improve negative symptoms and cognitive function in schizophrenia.Therefore, this study explore the efficacy of iTBS on negative symptoms and cognitive deficits in schizophrenia based on identifying the brain network connection of schizophrenia symptoms.

Firstly, we have used neuroimaging to find the left prefrontal cortex that is responsible for negative symptoms and cognitive function in schizophrenia. Then,we design this randomized double-blind sham-controlled clinical trial. Patients with schizophrenia will be randomly treated with iTBS or sham condition to the left dorsolateral prefrontal cortex(L-DLPFC) for continuous 10 days, theL-DLPFC will be targeted utilizing the localite neuronavigation system. The follow-ups are set at baseline, the 11th day and the 30th day after the end of treatment. The main outcome measures include the change in MCCB score, PANSS score, SANS score, SAPS score and the resting-state functional magnetic resonance imaging data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with schizophrenia in accordance with DSM-5
2. The disease duration ≤8 years
3. Received a steady dose of antipsychotic medication for least 4 weeks
4. The Global Deficit Score of MCCB ≥0.5 or the PANSS negative subscore ≥20
5. No obvious extrapyramidal side effects caused by antipsychotic drugs
6. Informed Consent

Exclusion Criteria:

1. Diagnosed with other mental disease in accordance with DSM-5
2. Combined with other severe physiological disease
3. Used antidepressants, mood stabilizer, or other psychoactive substances before
4. Drug or alcohol abuse
5. Pregnant or lactating
6. Contraindication to rTMS
7. Received rTMS or electroconvulsive therapy in the past 1 month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Change in MCCB | From baseline to 11days and the 30th day after the end of stimulation
  The MATRICS Consensus Cognitive Battery,It can be used for cognitive assessment of schizophrenia, bipolar disorder and other neuropsychiatric diseases,The MCCB covers nine cognitive domains including attention, information processing speed, verbal learning and memory, visual learning and memory, spatial working memory, reasoning, problem solving, social cognition, executive function and fine motor. The working memory domain does not include verbal working memory because the Chinese language would not make feasible the inclusion of the LNS test.
Change in Positive and Negative Symptm Scale(PANSS) score | From baseline to 11days and the 30th day after the end of stimulation
  The scale to assess the severity of symptoms in schizophrenia.It is an evaluation scale of 30 disparate items scored from 1 to 7 for psychopathological symptoms observed in patients presenting psychotic syndromes, especially schizophrenic states.Three scores obtained with this scale are generally calculated for evaluating three dimensions of the syndrome: positive, negative and general psychopathology, as part of a categorial or dimensional perspective.The minimum value is 30 points, and the maximum value is 210 points.The higher the score, the more severe the relevant symptom is.
Change in Scale for Assessment of Positive Symptoms(SAPS) score | From baseline to 11days and the 30th day after the end of stimulation
  This scale is used to assess the severity of positive symptoms in schizophrenia. Evaluating four dimensions of the positive symptoms including hallucination, delusion, strange behavior and disorders of the positive thinking form.There are 34 items in the scale, which are divided into four subscales and graded on a six-point scale. The total score of the scale is the sum of 34 individual items, reflecting the severity of positive symptoms. The score range is 0-170, the higher the score, the more severe the symptoms are. The total score of the comprehensive evaluation is the sum of the individual score of the overall evaluation item of the four subscales, which also reflects the severity of positive symptoms, the score range is 0-20. The comprehensive evaluation score of the subscale is the single score of the overall evaluation item of the four subscales, specifically reflecting the severity of the four dimensions of the positive symptoms, the score range is 0-5.
Change in Scale for Assessment of Negative Symptoms(SANS) score | From baseline to 11days and the 30th day after the end of stimulation
  This scale is used to assess the severity of negative symptoms in schizophrenia. Evaluating five dimensions of the negative symptoms including apathy, poverty of thought, abulia, social withdrawal and disorders of attention.There are 24 items in the scale, which are divided into five subscales and graded on a six-point scale. The total score of the scale is the sum of 24 individual items, reflecting the severity of positive symptoms. The score range is 0-120, the higher the score, the more severe the negative symptoms are. The total score of the comprehensive evaluation is the sum of the individual score of the overall evaluation item of the five subscales, which also reflects the severity of negative symptoms, the score range is 0-25. The comprehensive evaluation score of the subscale is the single score of the overall evaluation item of the five subscales, specifically reflecting the severity of the five dimensions of the negative symptoms, the score range is 0-5.
The data of resting-state functional magnetic resonance imaging | From baseline to 11days and the 30th day after the end of stimulation
  All patients undergo head MRI scans in Philips Achieva 3.0 T scanner and SIEMENS Prisma 3.0 T scanner.

SECONDARY OUTCOMES:
Change in Treatment Emergent Symptom Scale(TESS) score | From baseline to 11days and the 30th day after the end of stimulation
  The scale is used to assess the side effects of various psychotropic drugs in adult patients. Evaluation is based on patient statements, physical examination and laboratory results.The 34 symptoms were summarized into 6 groups of symptoms, including behavioral adverse reactions, laboratory tests, nervous system reactions, autonomic nervous system symptoms, cardiovascular system reactions and others.The scale evaluation requires a three-pronged assessment of each symptom: severity, the relationship between the symptom and the medication, and the treatment.
The blood sample | From baseline to 11days and the 30th day after the end of stimulation
  About 20ml blood samples were collected intravenously to test blood routine, liver and kidney function, electrolytes and other routine tests.

CONTACTS AND LOCATIONS:
Overall Officials: Renrong Wu, Prof, Principal Investigator — The Second Xiangya Hospital of Central South University Psychiatry Department
Locations (1):
- Second Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No